CLINICAL TRIAL: NCT06367231
Title: Serious Computer Games as a Proxy for Determining the Cognitive Status of Older Adults
Brief Title: SCGs as a Proxy for Determining the Cognitive Status of Older Adults
Status: Completed | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00134554
Record Dates: First submitted 2024-03-23; First posted 2024-04-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Mild Cognitive Impairment; Dementia; Alzheimer Disease; Healthy Aging; Cognitive Decline
Keywords: Serious computer game; computer games; VibrantMinds
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Serious Computer Game Intervention: Older Adults (healthy), Older adults with MCI, older adults with dementia
  Each participant will undergo three sessions, spaced one week apart. These sessions will take place either at locations that support the research team's activities or at the participants' homes, offering flexibility to accommodate individual circumstances. The format of these sessions can vary, being either group-based or individual.
  Each session is designed to last approximately one hour, with a maximum duration of 90 minutes to ensure thoroughness without overwhelming participants.
  Interventions: Other: VibrantMinds

INTERVENTIONS:
Other: VibrantMinds — We are exploring the potential of computer games to reveal insights into the cognitive abilities of older adults. We developed the VibrantMinds (https://vibrant-minds.org/vibrantminds2/start) platform, featuring five games: Whack-a-Mole, Bejeweled, Mahjong Solitaire, Word Search, and Memory Game. Our evaluation focused on the usability of these games, their appeal to users, and their effectiveness in enhancing cognitive functions. The next phase of our study aims to determine whether these games can offer meaningful data on the cognitive skills of older adults.
  Other Names: Serious Computer Games

SUMMARY:
Detecting memory problems early is crucial for treating conditions like Mild Cognitive Impairment (MCI), which often leads to dementia. Currently, doctors use tests in clinics to check for these issues. However, there's a growing need for better methods to monitor our cognitive skills over time. Computer games emerge as a cost-effective solution for assessing the brain functions of older adults.

In our study, we are investigating the potential of computer games to reflect the cognitive skills of older adults. We developed the VibrantMinds platform, featuring five games: Whack-a-Mole, Bejeweled, Mahjong Solitaire, Word Search, and Memory Game. We have evaluated these games for ease of use, enjoyment, and their impact on brain functions. Now, our goal is to determine whether these games can offer valuable insights into the cognitive skills of older adults.

We are collecting demographic data, game-playing data, and cognitive test results. Our analysis will determine the correlation between game data, cognitive test outcomes, and demographic information. Additionally, we will assess both the perceived and observed engagement of older adults as they play the games.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Calgary and/or Edmonton, Alberta, Canada
* sufficient English language skills to converse in English with research staff

Exclusion Criteria:

* Moderate or severe limitations in the control or movement of the upper extremity (e.g., severe arthritis, amyotrophic lateral sclerosis, multiple sclerosis)
* Visual and hearing impairments
* Attention deficit

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Older healthy adults (cognitively intact) Older adults with Mild Cognitive Impairment Older adults with Dementia
Sampling Method: Non-Probability Sample
Enrollment: 6 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Cognition - Global | At each session (3 sessions total, once per week, one week apart)
  The Montreal Cognitive Assessment (MoCA) is a brief 30-point test used to screen for cognitive dysfunction in areas including memory, language, visuospatial skills, executive functions, attention, concentration, and orientation. A score of 26 or above is considered normal. Lower scores suggest potential cognitive impairment.

SECONDARY OUTCOMES:
Cognition - Global | At each session (3 sessions total, once per week, one week apart)
  The Mini-Mental State Examination (MMSE) is a widely used 30-point questionnaire that assesses cognitive function, including orientation, recall, attention, calculation, language, and basic motor skills. A score of 24 or above typically indicates normal cognitive function, while lower scores suggest possible impairment.
Cognition - Executive Function | At each session (3 sessions total, once per week, one week apart)
  Trail Making Test, Part A and B. The norms and average completion times for the Trail Making Test (TMT) Parts A and B can vary significantly based on age, education, and the specific population being tested. However, general guidelines can provide some insight:
  TMT Part A: Average completion times for adults can range from 20 to 40 seconds. Younger adults and those with higher levels of education tend to complete Part A more quickly. Completion times increase with age.
  TMT Part B: This part is more complex and typically takes longer to complete, with average times ranging from 50 to 120 seconds.
Game Performance | Obtained during each game (game played at each session, once per week, one week apart)
  Level, Accuracy, Time
Game Engagement | At each session (3 sessions total, once per week, one week apart)
  Self-reported questionnaire of engagement and engagement indicators

CONTACTS AND LOCATIONS:
Locations (8):
- Canada (8):
  - Alzheimer Society of Alberta and Northwest Territories, Edmonton, Alberta
  - CapitalCare Corporate Services, Edmonton, Alberta
  - Edmonton Life Long Learners, Edmonton, Alberta
  - Institute for Continuing Care Education and Research, Edmonton, Alberta
  - Shepherd's Care Foundation, Edmonton, Alberta
  - St. Michael's Long Term Care Centre,, Edmonton, Alberta
  - Sherwood Care, Sherwood Park, Alberta
  - Tofield Health Centre, Tofield, Alberta

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: VibrantMinds Platform — https://vibrant-minds.org/vibrantminds2/start